CLINICAL TRIAL: NCT04787666
Title: Comparison of Non-invasive Methods of Lung Ventilation in Patients With Respiratory Failure in the Postoperative Period After Cardiac Surgery
Brief Title: Comparison of Non-invasive Methods of Lung Ventilation in Patients With Respiratory Failure After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Darya Ryabova, research worker, Russian national research center of surgery named after academian B. V. Petrovsky, Petrovsky National Research Centre of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01092005
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the first group: non-invasive mask ventilation (Experimental): Dinamika of the indicator p/F Ratio
  Interventions: Procedure: Using of non-invasive mask ventilation, high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) and non-invasive ventilation with a helmet
- the second group:high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) (Experimental): Dinamika of the indicator p/F Ratio
  Interventions: Procedure: Using of non-invasive mask ventilation, high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) and non-invasive ventilation with a helmet
- the third group:non-invasive ventilation with a helmet (Experimental): Dinamika of the indicator p/F Ratio
  Interventions: Procedure: Using of non-invasive mask ventilation, high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) and non-invasive ventilation with a helmet

INTERVENTIONS:
Procedure: Using of non-invasive mask ventilation, high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) and non-invasive ventilation with a helmet — Using of non-invasive mask ventilation, high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) and non-invasive ventilation with a helmet for tackling the problem of respiratory failure

SUMMARY:
Comparison of the effectiveness of three methods of non-invasive ventilation in patients with mild and moderate respiratory failure in the early postoperative period after cardiac surgery

DETAILED DESCRIPTION:
The study includes the comparison of the three methods of non-invasive ventilation: non-invasive mask ventilation, high-flow oxygen therapy through a nasal cannula (high-flow nasal oxygenation) and non-invasive ventilation with a helmet in patients with mild and moderate respiratory failure in the early postoperative period after cardiac surgery. It assumes 90 randomized patients:30 patients in three study groups male and female aged 30 to 60 years of age inclusive, with mild or moderate respiratory failure.The study will be randomized, single-center, prospective.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 30 years to 60 years inclusive
2. Decreased oxygenation function of the lungs (SpO2 less than 90%, PaO2/FiO2 less than 300, BH less than 25 per minute)
3. By data CT/x-ray examination of hypoventilation zones (pneumonia, atelectasis)
4. Consent the patient to participate in this study

Exclusion Criteria:

1. Tracheal intubation, absence of independent breathing
2. Unstable hemodynamics or hemodynamically significant rhythm disturbances
3. Acute violation of the cerebral blood supply
4. Shocks of various etiologies
5. Impossibility provide respiratory protection , high risk of aspiration
6. Lack of productive contact with the patient
7. Patient's refusal to participate in this study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 more than 300 | hospitalisation period, an average of 1 week
  Comparison of PaO2/FiO2 before/after research

SECONDARY OUTCOMES:
arterial blood oxygenation level | hospitalisation period, an average of 1 week
  Comparison arterial blood oxygenation level before/after research
maximum inspiratory volume | hospitalisation period, an average of 1 week
  Comparison maximum inspiratory volume before/after research

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A. Eremenko, prof, Study Director — Head of the Intensive Care Unit; Darya V. Ryabova, Principal Investigator — anesthesiologist-resuscitator
Locations (1):
- Petrovsky Research National Centre of Surgery, Moscow, Russia

REFERENCES:
- See also: The article — http://intensive-care.ru/index.php/acc/article/view/433/2685